CLINICAL TRIAL: NCT03659175
Title: Study on Clinical Features, Intestinal Flora and Standardized Treatment in Male Elderly With Small Intestinal Bacterial Overgrowth
Brief Title: Characteristic of Intestinal Flora in Male Elderly With Small Intestinal Bacterial Overgrowth
Acronym: IFOSIBO
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Ru Zhang MD, doctor of medcine, Chinese PLA General Hospital
Other Study IDs: RZhang
Record Dates: First submitted 2018-01-10; First posted 2018-09-06 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Small Intestinal Bacterial Overgrowth; Elderly; Male; 16s rRNA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — feces and intestinal biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- male elderly with SIBO: male elderly who was diagnosed as SIBO via 'lactulose breath test' (LBT). At the same time, they meet the following criteria:
  1. no use of antibiotics in the past 1 month.
  2. no use of prokinetic drugs and probiotics in the past 1 week.
  3. without these diseases: active inflammation, cardiac insufficiency, respiratory insufficiency, hepatic insufficiency, renal insufficiency, cirrhosis, thyroid diseases, Crohn disease, ulcerative colitis, hepatobiliary and pancreatic disease.
  Interventions: Other: SIBO
- male elderly without SIBO: male elderly without SIBO after 'lactulose breath test'. At the same time, they meet the following criteria:
  1. no use of antibiotics in the past 1 month.
  2. no use of prokinetic drugs and probiotics in the past 1 week.
  3. without these diseases: active inflammation, cardiac insufficiency, respiratory insufficiency, hepatic insufficiency, renal insufficiency, cirrhosis, thyroid diseases, Crohn disease, ulcerative colitis, hepatobiliary and pancreatic disease.

INTERVENTIONS:
Other: SIBO — SIBO: Small intestinal bacterial overgrowth, refers to a bacterial overgrowth due to organic or functional stasis in small intestine, leading to the change in number or types of bacteria in small intestine.
  Groups: male elderly with SIBO

SUMMARY:
We will focus on the intestinal flora structure, risk factors and clinical features of male elderly with SIBO in our study.

DETAILED DESCRIPTION:
Our previous study had found that the prevalence rate of small intestinal bacterial overgrowth(SIBO) in male elderly was high up to 63.1%. In the recent years, SIBO has been found be associated not only with abdominal symptoms such as abdominal distention, pain and so on, but also with various diseases such as diabetes, Alzheimer's disease, joint pain, chronic prostatitis, fatty liver, liver cirrhosis etc. SIBO has significant impact on the health of elderly. Methane and hydrogen lactulose breath test(LBT) is effective and noninvasive for the diagnosis of SIBO. High throughput sequencing is a leading technique for the study of intestinal microflora.

Although more and more studies have focused their concern on the intestinal flora now, few SIBO-related studies are available in elderly patients. But we have found SIBO was very popular in the elderly. The conflict between high prevalence rate of SIBO in elderly and very few relevant studies is barrier to study of pathophysiology, early diagnosis and treatment of SIBO in elderly adults.

So in our study, we will apply LBT and high throughput sequencing technique to study the intestinal flora structure, risk factors and clinical features of male elderly patients with SIBO. And further, we will try to develop standard treatment for elderly patients with SIBO.

ELIGIBILITY:
Inclusion Criteria:

* no use of antibiotics in the past 1 month, no use of prokinetic drugs and probiotics in the past 1 week

Exclusion Criteria:

* active inflammation, cardiac insufficiency, respiratory insufficiency, hepatic insufficiency, renal insufficiency, cirrhosis, thyroid diseases, Crohn disease, ulcerative colitis, hepatobiliary and pancreatic disease

Ages: 65 Years to 98 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — male
Study Population: male elderly outpatients at Department of Gastroenterology, Nanlou Division, Chinese PLA General Hospita, Beijing, China
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-10-15 (Estimated); Primary Completion 2019-12-10 (Estimated); Study Completion 2020-05-10 (Estimated)

PRIMARY OUTCOMES:
amplicon sequencing of intestinal microflora | 1 year
  We will collect specimen(include feces and intestinal biopsy), then amplicon sequencing of intestinal microflora in specimen. And study the difference in intestinal microflora structure bwteen male elderly with and without SIBO.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Wan, Study Director — Director
Locations (1):
- Chinese PLA general hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
the data of these male elederly enrolled in the study are secret on account of their status